CLINICAL TRIAL: NCT01681875
Title: Project 1, Study 1: Investigating the Impact of Nicotine Using Spectrum Cigarettes
Acronym: P1S1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Masonic Cancer Center, University of Minnesota (Other); Brown University (Other); Johns Hopkins University (Other); University of California, San Francisco (Other); M.D. Anderson Cancer Center (Other); University of Pennsylvania (Other); Duke University (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: U54DA031659 (NIH); U54DA031659-01 (NIH)
Record Dates: First submitted 2012-08-30; First posted 2012-09-10 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Tobacco Dependence
Keywords: Biomarkers of exposure; Compensatory smoking; Nicotine dependence; Reduced nicotine cigarettes; Tobacco withdrawal
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 0.8 mg nicotine with 9 mg tar (Experimental): very low nicotine content cigarettes
  SPECTRUM Cigarette: 0.8 (±0.15) mg nicotine with 9 (±1.5) mg tar (standard nicotine and tar yields of commercially-available cigarettes; control condition)
  Interventions: Other: very low nicotine content cigarettes
- 0.26 mg nicotine with 9 mg tar (Experimental): very low nicotine content cigarettes
  SPECTRUM Cigarette: 0.26 (±0.06) mg nicotine with 9 (±1.5) mg tar
  Interventions: Other: very low nicotine content cigarettes
- 0.12 mg nicotine with 9 mg tar (Experimental): very low nicotine content cigarettes
  SPECTRUM Cigarette: 0.12 (±0.03) mg nicotine with 9 (±1.5) mg tar
  Interventions: Other: very low nicotine content cigarettes
- 0.07 mg nicotine with 9 mg tar (Experimental): very low nicotine content cigarettes
  SPECTRUM Cigarette: 0.07 (±0.02) mg nicotine with 9 (±1.5) mg tar
  Interventions: Other: very low nicotine content cigarettes
- 0.03 mg nicotine with 9 mg tar (Experimental): very low nicotine content cigarettes
  SPECTRUM Cigarette: 0.03 (±0.01) mg nicotine with 9 (±1.5) mg tar
  Interventions: Other: very low nicotine content cigarettes
- 0.04 mg nicotine with 13 mg tar (Experimental): very low nicotine content cigarettes
  SPECTRUM Cigarette: 0.04 (±0.02) mg nicotine with 13 (±2) mg tar
  Interventions: Other: very low nicotine content cigarettes
- Usual brand (Other): very low nicotine content cigarettes
  Usual brand cigarettes (control condition)
  Interventions: Other: very low nicotine content cigarettes

INTERVENTIONS:
Other: very low nicotine content cigarettes

SUMMARY:
Project 1, Study 1 will evaluate the relationship between nicotine yield of very low nicotine content cigarettes and cigarettes smoked per day, nicotine exposure, discomfort/dysfunction, other health-related behaviors, nicotine/tobacco dependence, biomarkers of tobacco exposure, intention to quit, compensatory smoking, other tobacco use, cigarette characteristics, cognitive function, cardiovascular function, and perceived risk. We will also consider differences between conditions in compliance with product use.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Smoke an average of at least five cigarettes per day for at least 1 year
* Breath CO levels > 8 ppm (if ≤ 8 ppm, then NicAlert Strip > 2)

Exclusion Criteria:

* Intention to quit smoking in the next 30 days
* Currently seeking treatment for smoking cessation
* Currently using nicotine replacement therapies or other pharmacotherapies as cessation aid (intermittent use acceptable)
* A quit attempt in the past 30 days resulting in greater than 3 days of abstinence
* Using other tobacco products more than 9 days in the past 30 days
* Significant unstable medical conditions (Any significant change in a serious medical condition occurring during the past 3 months including, cardiovascular disease, COPD, and cancer, as determined by the licensed medical professional at each site)
* Significant unstable psychiatric conditions (Any significant change in psychiatric symptoms during the past 3 months as determined by the licensed medical professional at each site)
* Schizophrenia and schizoaffective disorder
* Psychiatric medication changes in the past 3 months
* Positive toxicology screen for any of the following drugs: cocaine, opiates, methadone, benzodiazepines, barbiturates, amphetamines, methamphetamines, and PCP

  1. Marijuana will be tested for but will not be an exclusionary criterion.
  2. Participants with valid prescriptions for opiates, benzodiazepines, barbiturates, amphetamines or methadone will not be excluded.
  3. Participants failing the toxicology screen will be allowed to re-screen once.
* Blood alcohol level > 0.01

  a. Participants failing the blood alcohol screen will be allowed to re-screen once.
* Binge drinking alcohol (more than 9 days in the past 30 days, 4/5 in a 2 hour period(female/male))
* Pregnant or breastfeeding
* Smoking 'roll your own cigarettes' exclusively
* Currently taking anticonvulsant medication
* CO reading >80 ppm
* Systolic BP greater than or equal to 160

  a. Participants failing for blood pressure will be allowed to re-screen once.
* Diastolic BP greater than or equal to 100

  a. Participants failing for blood pressure will be allowed to re-screen once.
* Systolic BP below 90

  a. Participants failing for blood pressure will be allowed to re-screen once.
* Diastolic BP below 50

  a. Participants failing for blood pressure will be allowed to re-screen once.
* Heart rate greater than or equal to 115bpm

  a. Participants failing for heart rate will be allowed to re-screen once.
* Heart rate lower than 45bpm

  a. Participants failing for heart rate will be allowed to re-screen once.
* Indicating any suicidal ideation in the past month or suicide attempts in the past 10 years
* Inability to independently read and comprehend the consent form and other written study materials and measures
* Having participated in a research study during the past three months in which the participant:

  1. Smoked a cigarette that was not his/her usual brand cigarette for more than one day
  2. Used any tobacco products beyond normal use for more than one day
  3. Used any nicotine replacement products or smoking cessation medications for more than one day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of cigarettes smoked per day | End of 6 week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Donny, PhD, Study Director — University of Pittsburgh
Locations (9):
- United States (9):
  - University of California San Francisco, San Francisco, California
  - Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota Medical School Duluth, Duluth, Minnesota
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island

REFERENCES:
- [Background] Donny EC, Jones M. Prolonged exposure to denicotinized cigarettes with or without transdermal nicotine. Drug Alcohol Depend. 2009 Sep 1;104(1-2):23-33. doi: 10.1016/j.drugalcdep.2009.01.021. Epub 2009 May 15. PMID 19446968
- [Background] Hatsukami DK, Kotlyar M, Hertsgaard LA, Zhang Y, Carmella SG, Jensen JA, Allen SS, Shields PG, Murphy SE, Stepanov I, Hecht SS. Reduced nicotine content cigarettes: effects on toxicant exposure, dependence and cessation. Addiction. 2010 Feb;105(2):343-55. doi: 10.1111/j.1360-0443.2009.02780.x. PMID 20078491
- [Background] Benowitz NL, Dains KM, Hall SM, Stewart S, Wilson M, Dempsey D, Jacob P 3rd. Smoking behavior and exposure to tobacco toxicants during 6 months of smoking progressively reduced nicotine content cigarettes. Cancer Epidemiol Biomarkers Prev. 2012 May;21(5):761-9. doi: 10.1158/1055-9965.EPI-11-0644. Epub 2012 Feb 21. PMID 22354905
- [Background] Donny EC, Houtsmuller E, Stitzer ML. Smoking in the absence of nicotine: behavioral, subjective and physiological effects over 11 days. Addiction. 2007 Feb;102(2):324-34. doi: 10.1111/j.1360-0443.2006.01670.x. PMID 17222288
- [Derived] Denlinger-Apte RL, Tidey JW, Koopmeiners JS, Hatsukami DK, Smith TT, Pacek LR, McClernon FJ, Donny EC. Correlates of support for a nicotine-reduction policy in smokers with 6-week exposure to very low nicotine cigarettes. Tob Control. 2019 May;28(3):352-355. doi: 10.1136/tobaccocontrol-2018-054622. Epub 2018 Nov 1. PMID 30385649
- [Derived] Dermody SS, McClernon FJ, Benowitz N, Luo X, Tidey JW, Smith TT, Vandrey R, Hatsukami D, Donny EC. Effects of reduced nicotine content cigarettes on individual withdrawal symptoms over time and during abstinence. Exp Clin Psychopharmacol. 2018 Jun;26(3):223-232. doi: 10.1037/pha0000179. Epub 2018 Mar 5. PMID 29504780
- [Derived] Rupprecht LE, Koopmeiners JS, Dermody SS, Oliver JA, al'Absi M, Benowitz NL, Denlinger-Apte R, Drobes DJ, Hatsukami D, McClernon FJ, Pacek LR, Smith TT, Sved AF, Tidey J, Vandrey R, Donny EC. Reducing nicotine exposure results in weight gain in smokers randomised to very low nicotine content cigarettes. Tob Control. 2017 Mar;26(e1):e43-e48. doi: 10.1136/tobaccocontrol-2016-053301. Epub 2016 Nov 17. PMID 27856940
- [Derived] Dermody SS, Tidey JW, Denlinger RL, Pacek LR, al'Absi M, Drobes DJ, Hatsukami DK, Vandrey R, Donny EC. The Impact of Smoking Very Low Nicotine Content Cigarettes on Alcohol Use. Alcohol Clin Exp Res. 2016 Mar;40(3):606-15. doi: 10.1111/acer.12980. Epub 2016 Feb 25. PMID 26916879
- [Derived] Donny EC, Denlinger RL, Tidey JW, Koopmeiners JS, Benowitz NL, Vandrey RG, al'Absi M, Carmella SG, Cinciripini PM, Dermody SS, Drobes DJ, Hecht SS, Jensen J, Lane T, Le CT, McClernon FJ, Montoya ID, Murphy SE, Robinson JD, Stitzer ML, Strasser AA, Tindle H, Hatsukami DK. Randomized Trial of Reduced-Nicotine Standards for Cigarettes. N Engl J Med. 2015 Oct;373(14):1340-9. doi: 10.1056/NEJMsa1502403. PMID 26422724